CLINICAL TRIAL: NCT04741906
Title: Outcome of Dental Implant Therapy in Patients Treated With Antiresorptive Medication
Status: Recruiting | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Amgen (Industry); Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Sanne Werner Moeller Andersen, Oral and Maxillofacial Surgeon, Copenhagen University Hospital at Herlev
Other Study IDs: Oral rehabilitation of MRONJ
Record Dates: First submitted 2021-01-21; First posted 2021-02-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Missing Teeth; Implants; Cancer; Osteoporosis
Keywords: Dental implants; High dose antiresorptive medication; Rehabilitation; Denosumab; Bisphosphonate; Oral rehabilitation; Adjuvant dose antiresorptive medication; Low dose antiresorptive medication; Bone modifying agents
MeSH Terms: conditions — Anodontia; Neoplasms; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Patient with osteoporosis - antiresorptive treatment > 4 years. Previous tooth extraction: Patient with osteoporosis - antiresorptive treatment > 4 years who have had previous tooth extraction without development of MRONJ
  Interventions: Procedure: Dental implant surgery; Procedure: Prosthetic treatment
- Patient with osteoporosis - antiresorptive treatment > 4 years. Previous resection: Patient with osteoporosis - antiresorptive treatment > 4 years who have lost teeth due to having previous osteonecrosis of the jaw which has been successfully surgically treated and healed for at least 3 months without recurrence
  Interventions: Procedure: Dental implant surgery; Procedure: Prosthetic treatment
- Patient with osteoporosis - antiresorptive treatment > 4 years. Simultaneously with resection: Patient with osteoporosis - antiresorptive treatment > 4 years with ongoing osteonecrosis of the jaw to be surgically treated with block resection of the lower jaw and insertion of a titanium reconstruction plate. Simultaneous insertion of dental implants, or resection of the upper jaw where there is sufficient remaining bone volume to have implants inserted simultaneously (without bone augmentation)
  Interventions: Procedure: Dental implant surgery; Procedure: Prosthetic treatment
- Patient with cancer - adjuvant dose antiresorptive treatment. Previous tooth extraction: Patient with cancer (breast, prostate or multiple myeloma) - adjuvant dose antiresorptive treatment who have had previous tooth extraction without development of MRONJ
  Interventions: Procedure: Dental implant surgery; Procedure: Prosthetic treatment
- Patient with cancer - adjuvant dose antiresorptive treatment. Previous resection: Patient with cancer (breast, prostate or multiple myeloma) - adjuvant dose antiresorptive treatment who have lost teeth due to having previous osteonecrosis of the jaw which has been successfully surgically treated and healed for at least 3 months without recurrence
  Interventions: Procedure: Dental implant surgery; Procedure: Prosthetic treatment
- Patient with cancer - adjuvant dose antiresorptive treatment. Simultaneously with resection: Patient with cancer (breast, prostate or multiple myeloma) - adjuvant dose antiresorptive treatment with ongoing osteonecrosis of the jaw to be surgically treated with block resection of the lower jaw and insertion of a titanium reconstruction plate. Simultaneous insertion of dental implants, or resection of the upper jaw where there is sufficient remaining bone volume to have implants inserted simultaneously (without bone augmentation)
  Interventions: Procedure: Dental implant surgery; Procedure: Prosthetic treatment
- Cancer patient treated with high dose antiresorptive treatment. Previous tooth extraction: Cancer patient treated with high dose antiresorptive treatment who have had previous tooth extraction without development of MRONJ
  Interventions: Procedure: Dental implant surgery; Procedure: Prosthetic treatment
- Cancer patient treated with high dose antiresorptive treatment. Previous resection: Cancer patient treated with high dose antiresorptive treatment who have lost teeth due to having previous osteonecrosis of the jaw which has been successfully surgically treated and healed for at least 3 months without recurrence
  Interventions: Procedure: Dental implant surgery; Procedure: Prosthetic treatment
- Cancer patient treated with high dose antiresorptive treatment. Simultaneously with resection: Cancer patients (breast, prostate or multiple myeloma) treated with high dose antiresorptive treatment with ongoing osteonecrosis of the jaw to be surgically treated with block resection of the lower jaw and insertion of a titanium reconstruction plate. Simultaneous insertion of dental implants, or resection of the upper jaw where there is sufficient remaining bone volume to have implants inserted simultaneously (without bone augmentation)
  Interventions: Procedure: Dental implant surgery; Procedure: Prosthetic treatment

INTERVENTIONS:
Procedure: Dental implant surgery — Dental surgery in patients treated with antiresorptive medication
Procedure: Prosthetic treatment — Prosthetic treatment and loading of the dental implants

SUMMARY:
Aim of the study is to examine the feasibility of dental implant insertion in patients receiving high, adjuvant and low dose > 4 years.

DETAILED DESCRIPTION:
The hypothesis of the present study is that dental implant therapy using submerged healing is feasible and predictable in patients receiving high, adjuvant or low dose AR for more than 4 years, as documented by clinical and radiographic signs of osseointegration after 3-4 months, sufficient implant stability for abutment connection, and implant survival rates comparable to those of healthy individuals after one year of prosthetic loading.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cancer or osteoporosis, treated with antiresorptive treatment.
* The patients should have sufficient compliance, this includes willingness to have the planned assessments
* The patient should have an expected life span at enrollment of at least 2 years.
* The local bone quality and quantity should be sufficient for implant insertion without bone augmentation and is classified according to the classification by Cawood & Howell 1988.

Exclusion Criteria:

* > 10 cigarettes daily
* HbA1c > 53 mmol/mol
* Poor oral hygiene
* Poor general condition: ECOG score 3 or 4.
* Poor prognosis: Expected survival <2 year is an exclusion cause.
* Presence of metastases of the liver brain.
* Poor local jaw bone quality acc. to Cawood classification stage 3 or 4.
* Unwillingness to comply with the planned assessments and recordings

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Total or partial toothless patients treated with antiresorptive medication, treated at Copenhagen University Hospital due to treatment with high dose, adjuvant, or low dose > 4 years, antiresorptive treatment. The patients had former tooth extractions or resections of the jaw at our clinic.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dental implant survival | 3 months
  Defined as presence of the implant in the jaw after initial implant surgery before abutment surgery
Dental implant survival | 6 months
  Defined as presence of the implant at time of final prosthetics
Dental implant survival | 18 months
  Defined as presence of the implant 1 year after loading of the final prosthetics
Dental implant survival | 30 months
  Defined as presence of the implant 2 years after loading of the final prosthetics
Dental Implant success | 30 months
  Defined as less marginal bone loss than 1.5 mm the first year, and 0.2 mm per year thereafter at time of assessment
Absence of medical related osteonecrosis of the jaw (MRONJ) | 30 months
  Defined as no exposed bone, no fistula, no radiologic sign of MRONJ

SECONDARY OUTCOMES:
Oral Health Impact Profile | 30 months
  Using OHIP-14 questionnaire to evaluate oral health-related quality of life
EORTC QLQ-H&N 35 | 30 months
  Performance of the EORTC questionnaire for the assessment of quality of life in head and neck cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Sanne Werner Moeller Andersen, DDS, Principal Investigator — Copenhagen University Hospital, Maxillofacial surgery
Locations (1):
- Copenhagen University Hospital, Maxillofacial Department, Copenhagen, Danmark, Denmark

REFERENCES:
- [Derived] Ottesen C, Andersen SWM, Jensen SS, Kofod T, Gotfredsen K. Medication-related osteonecrosis of the jaw and successful implant treatment in a patient on high-dose antiresorptive medication: A case report. Clin Exp Dent Res. 2022 Oct;8(5):1059-1067. doi: 10.1002/cre2.620. Epub 2022 Jul 27. PMID 35894761
- [Derived] Andersen SWM, Ottesen C, Gotfredsen K, Jensen SS, Kofod T, Schiodt M. Outcome of healing after dental implant placement in patients with cancer on high-dose antiresorptive medications: a prospective feasibility study. Oral Maxillofac Surg. 2023 Mar;27(1):89-100. doi: 10.1007/s10006-022-01042-5. Epub 2022 Jan 27. PMID 35084584